CLINICAL TRIAL: NCT01635166
Title: A Multi-centre, Prospective, Uncontrolled Post Market Clinical Follow-up Study (PMCFS) to Monitor the Survival and Performance of the DeltaMotion Cup System in Subjects Requiring a Total Hip Replacement
Brief Title: Multi-centre Study to Assess the Long-term Performance of the Deltamotion Cup System in Primary Hip Replacement Surgery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: DePuy International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT11/01
Record Dates: First submitted 2012-02-06; First posted 2012-07-09 (Estimated); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Rheumatoid Arthritis; Osteoarthritis; Post-traumatic Arthritis; Avascular Necrosis; Traumatic Femoral Fractures; Congenital Hip Dysplasia
Keywords: Arthroplasty; Replacement; Hip; Cementless; Ceramic on Ceramic
MeSH Terms: conditions — Arthritis, Rheumatoid; Osteoarthritis; Osteonecrosis; Hip Dislocation, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Delta Motion (Other): A cementless acetabular cup with a pre-assembled ceramic liner for use in total hip replacement
  Interventions: Device: Delta Motion

INTERVENTIONS:
Device: Delta Motion — A cementless acetabular cup with a pre-assembled ceramic liner for use in total hip replacement.

SUMMARY:
The purpose of this study is to monitor the performance of the DeltaMotion cup system in the treatment of patients with hip joint disease requiring a total hip replacement.Patients who enter the study will be evaluated at regular intervals following hip surgery using patient, clinical and x-ray assessments.

ELIGIBILITY:
Inclusion Criteria

i) Male or female subjects, aged between 18 and 70 years inclusive.

ii) Subjects who are able to give voluntary, written informed consent to participate in this Clinical Investigation and from whom consent has been obtained.

iii) Subjects who, in the opinion of the Investigator, are able to understand this Clinical Investigation, co-operate with the investigational procedures and are willing to return to the hospital for all the required post-operative follow-ups.

iv) Subjects suitable for a cementless total hip replacement using the DeltaMotion Cup System, in accordance with all applicable Instructions For Use

Exclusion Criteria

i) Subjects who, in the opinion of the Investigator, have an existing condition that would compromise their participation and follow-up in this Clinical Investigation.

ii) Women who are pregnant.

iii) Subjects who are known drug or alcohol abusers or with psychological disorders that could affect follow-up care or treatment outcomes.

iv) Subjects who have participated in a Clinical Investigation with an investigational product in the last 12 months.

v) Subjects who are currently involved in any injury litigation claims.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2012-07-01 (Actual); Primary Completion 2018-02-08 (Actual); Study Completion 2018-02-08 (Actual)

PRIMARY OUTCOMES:
Kaplan-Meier survivorship | 3 years
  To determine survivorship of the DeltaMotion Cup System at 3 years

SECONDARY OUTCOMES:
Kaplan-Meier survivorship | 10yrs post-surgery
  To determine survivorship of the DeltaMotion Cup System at 10 years
Harris Hip Score | 10yrs post-surgery
  Change from baseline in the Harris Hip Score. The Harris Hip Score is used to measure the outcome of total hip replacement and covers the areas of pain, function, absence of deformity and range of motion.
Oxford Hip Score | 10yrs post-surgery
  Change from baseline in the Oxford Hip Score. The Oxford hip score is a patient completed outcomes score which is designed to assess function and pain with patients undergoing hip replacement surgery.
University of California Los Angeles (UCLA) Score | 10yrs post-surgery
  Change from baseline in the UCLA Quality of Life Score. UCLA is a patient completed outcome score used in hip replacement
Western Ontario and McMaster Universities (WOMAC) Score | 10yrs post-surgery
  Change from baseline in the WOMAC. WOMAC is a patient complete outcome score to assess pain, disability and joint stiffness in Osteoarthritis of the hip and knee
Radiological analysis | 10yrs post-surgery
  * Acetabular Migration (vertical or horizontal) less than 5mm
  * Acetabular Migration (varus or valgus) less than 5 degrees
  * No loosening - absence of acetabular radiolucencies of greater than 2mm in two zones.

CONTACTS AND LOCATIONS:
Locations (3):
- India (2):
  - Apollo Speciality hospital, 320 Anna Salai, Chennai
  - All India Institute of Medical Sciences, Ansari nagar, South Extension, New Dehli
- Robert Jones and Agnes Hunt, Oswestry, United Kingdom